CLINICAL TRIAL: NCT04839107
Title: Institutional COVID-19 Patient Registry
Brief Title: Institutional Registry on Outpatient and Hospitalized COVID-19 Infected Patients
Acronym: IRCIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 5604
Record Dates: First submitted 2021-01-29; First posted 2021-04-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Creation of an Institutional Registry system for patients with confirmed COVID-19 infection with the collection of epidemiological data, risk factors, diagnosis, prognoses, treatment, follow-up and survival.

DETAILED DESCRIPTION:
Ambispective observational cohort with administrative admission date corresponding to the day of positivity of the PCR test for COVID-19, and discharge date of the cohort to the date corresponding to the epidemiological discharge, last contact with the health system and / or date of death.

Due to its institutional nature, the registry will collect data from the different patients who are assisted at different levels of the institution: emergency department, hospitalization in the general ward, critical areas, outpatient monitoring (including telemedicine) and home hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient assisted by HIBA adult services
* Patient diagnosed with COVID-19

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with COVID-19, evaluated and followed in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | From the date of the positivization of the PCR to the date of death or epidemiological discharge, whichever occurs first, assessed up to 30 days.
  Proportion of deceased persons from PCR positivity to epidemiological status out of the total number of infected persons followed in the same period
Readmission rate | Within a month of discharge
  Requirements for re-admission during the post-discharge period for a COVID hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano, CABA, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No